CLINICAL TRIAL: NCT03659136
Title: XENERA™1: A Multi-centre, Double-blind, Placebo-controlled, Randomised Phase II Trial to Compare Efficacy of Xentuzumab in Combination With Everolimus and Exemestane Versus Everolimus and Exemestane in Women With HR+ / HER2- Metastatic Breast Cancer and Non-visceral Disease
Brief Title: The XENERA™ 1 Study Tests Xentuzumab in Combination With Everolimus and Exemestane in Women With Hormone Receptor Positive and HER2-negative Breast Cancer That Has Spread
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1280-0022; 2017-003131-11 (EudraCT Number)
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Results first posted 2022-09-29 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — xentuzumab; Everolimus; exemestane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Xentuzumab/everolimus/exemestane (Experimental)
  Interventions: Drug: Xentuzumab; Drug: Everolimus; Drug: Exemestane
- Placebo/everolimus/exemestane (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Everolimus; Drug: Exemestane

INTERVENTIONS:
Drug: Xentuzumab — Intravenous infusion
  Arms: Xentuzumab/everolimus/exemestane
Drug: Placebo — Intravenous infusion
  Arms: Placebo/everolimus/exemestane
Drug: Everolimus — Tablet
Drug: Exemestane — Tablet

SUMMARY:
The main objective of the trial is to assess the efficacy of xentuzumab in combination with everolimus and exemestane over everolimus and exemestane in patients with HR+/ HER2- advanced or metastatic breast cancer and non-visceral disease.

ELIGIBILITY:
Inclusion Criteria:

* Documented histologically confirmed breast cancer with ERand/ or PgR-positive and HER2-negative status
* Locally advanced or metastatic breast cancer not deemed amenable to curative surgery or curative radiation therapy
* Archival tumour sample available at the time of informed consent and provided to the central laboratory around the time of randomisation. Patients must provide a formalin-fixed paraffin embedded (FFPE) tissue biopsy sample preferably taken at the time of presentation with recurrent or metastatic disease (provision of a biopsy sample taken from the bone is not acceptable).
* Patients must satisfy the following criteria for prior therapy:

  * Disease progression during treatment or within 12 months of completion of endocrine adjuvant therapy or
  * Disease progression while on or within 1 month after the end of prior endocrine therapy for advanced/metastatic breast cancer (Note: the endocrine therapy does not have to be the treatment immediately prior to trial entry).
* Patients must have

  * At least one measurable non-visceral lesion according to RECIST version 1.1 in either lymph nodes, soft tissue, skin and/or
  * At least one measurable non-visceral lesion according to RECIST version 1.1 as lytic or mixed (lytic + blastic) in bone and/or
  * At least one non-measurable (lytic, mixed lytic + blastic, or blastic) bone lesion according to RECIST version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1.
* Fasting glucose <8.9 mmol/L (<160 mg/dL) and HbA1c <8.0%
* Adequate organ function

Exclusion Criteria:

* Previous treatment with agents targeting the IGF pathway, AKT, or mTOR pathways
* Prior treatment with exemestane (except adjuvant exemestane stopped >12 months prior to start of study treatment as long as the patient did not recur during or within 12 months after the end of adjuvant exemestane)
* Evidence of visceral metastasis/es (i.e. liver, lung, peritoneal, pleural metastases, malignant pleural effusions, malignant peritoneal effusions) at screening. NOTE: Patients with a past history of visceral metastases are eligible if visceral metastases have completely resolved at least 3 months
* History or evidence of metastatic disease to the brain
* Leptomeningeal carcinomatosis
* More than 1 prior line of chemotherapy for HR+ HER2- metastatic breast cancer
* Radiotherapy within 4 weeks prior to the start of study treatment
* Use of concomitant systemic sex hormone therapy
* History or presence of cardiovascular abnormalities
* Known pre-existing interstitial lung disease
* Further exclusion criteria apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (16):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Cancer Treatment Centers of America at Western Regional Medical Center, Goodyear, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - University of California San Francisco, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - Florida Cancer Specialists, Fort Myers, Florida
  - University Cancer and Blood Center, Athens, Georgia
  - Hematology Oncology of Indiana, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - HCA MidAmerica Division, Inc., Kansas City, Missouri
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Southwestern Regional Medical Center, Tulsa, Oklahoma
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Utah Cancer Specialists Cancer Center, Salt Lake City, Utah
  - Northwest Medical Specialties, PLLC, Tacoma, Washington
- Australia (2):
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Peninsula Haematology & Oncology, Frankston, Victoria
- Belgium (4):
  - Brussels - UNIV Saint-Luc, Brussels
  - Brussels - UNIV UZ Brussel, Jette
  - Kortrijk - HOSP AZ Groeninge Kennedylaan, Kortrijk
  - UZ Leuven, Leuven
- CHU de Quebec-Universite Laval Research Centre, Québec, Canada
- France (7):
  - INS Sainte Catherine, Avignon
  - HOP Victor Hugo, Le Mans
  - INS Paoli-Calmettes, Marseille
  - INS Curie, Paris
  - HOP Européen G. Pompidou, Paris
  - HOP Lyon Sud, Pierre-Bénite
  - INS Claudius Regaud IUCT-Oncopole, Toulouse
- Germany (2):
  - Universitätsklinikum Erlangen, Erlangen
  - Vincentius-Diakonissen-Kliniken gAG, Karlsruhe
- Greece (5):
  - General Hospital of Athens "Alexandra", Athens
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Larisa, Oncology Clinic, Larissa
  - Metropolitan Hospital, Oncology Clinic, Neo Faliro, Athens
  - Euromedica Kyanous Stavros General Hospital, Thessaloniki
- Italy (3):
  - Istituto Nazionale IRCCS Tumori Fondazione Pascale, Napoli
  - Iov, Irccs, Padua
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
- Portugal (3):
  - Fundação Champalimaud,, Lisbon
  - Hospital Beatriz Ângelo, Loures
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Spain (10):
  - Hospital Teresa Herrera, A Coruña
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Instituto Valenciano de Oncología, Valencia
  - Clínica Quirón de Valencia, Valencia
  - Hospital Clínico de Valencia, Valencia
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Schmid P, Cortes J, Joaquim A, Janez NM, Morales S, Diaz-Redondo T, Blau S, Neven P, Lemieux J, Garcia-Saenz JA, Hart L, Biyukov T, Baktash N, Massey D, Burris HA 3rd, Rugo HS. XENERA-1: a randomised double-blind Phase II trial of xentuzumab in combination with everolimus and exemestane versus everolimus and exemestane in patients with hormone receptor-positive/HER2-negative metastatic breast cancer and non-visceral disease. Breast Cancer Res. 2023 Jun 12;25(1):67. doi: 10.1186/s13058-023-01649-w. PMID 37308971
- [Derived] Schmid P, Sablin MP, Bergh J, Im SA, Lu YS, Martinez N, Neven P, Lee KS, Morales S, Perez-Fidalgo JA, Adamson D, Goncalves A, Prat A, Jerusalem G, Schlieker L, Espadero RM, Bogenrieder T, Huang DC, Crown J, Cortes J. A phase Ib/II study of xentuzumab, an IGF-neutralising antibody, combined with exemestane and everolimus in hormone receptor-positive, HER2-negative locally advanced/metastatic breast cancer. Breast Cancer Res. 2021 Jan 15;23(1):8. doi: 10.1186/s13058-020-01382-8. PMID 33451345
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-centre, double-blind, placebo-controlled, randomised trial which assess the efficacy of of xentuzumab in combination with everolimus and exemestane over everolimus and exemestane in patients with Hormon Receptor+ (HR+)/ Human epidermal growth factor receptor 2 (HER2)- advanced or metastatic breast cancer and non-visceral disease.
Pre-assignment Details: All patients were screened for eligibility prior to participation in the trial. Patients were screened from 53 investigational sites in 11 countries, to ensure that they (the patients) strictly met all inclusion and none of the exclusion criteria. Screening could occur 1-28 days prior to randomisation to study treatment, patients were not to be randomised if any of the entry criteria were violated. Re-screening was allowed but only once per patient.
Groups:
- 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane: 1000 mg concentrate for solution for infusion of Xentuzumab (BI 836845) (10mg/mL supplied in 20mL vials (200mg/vial)) was administered once weekly as intravenous infusion over 1 hour on day 1, 8, 15 and 22 of 28-days cycles and on day 1, 8, 15, 22, 29, 36, 43 and 50 of 56-day cycles and tablets of 10 mg of Everolimus (Afinitor®) and tablets of 25 mg Exemestane (Aromasin®) were administered orally once per day at approximately the same time of day, after a meal.
- Placebo + 10 mg Everolimus + 25 mg Exemestane: Concentrate for solution for infusion of Placebo was administered once weekly as intravenous infusion of 1 hour on day 1, 8, 15 and 22 of 28-days cycles and on day 1, 8, 15, 22, 29, 36, 43 and 50 of 56-day cycles and tablets of 10 mg of Everolimus (Afinitor®) and tablets of 25 mg Exemestane (Aromasin®) were administered orally once per day at approximately the same time of day, after a meal.
Period: Overall Study
Arm/Group | 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane | Placebo + 10 mg Everolimus + 25 mg Exemestane
Started (Randomised) | 52 | 51
Treated | 50 | 51
On-treatment at Cut-off Date for Primary Analysis | 9 | 12
Completed (Completed = Number of participants on treatment at the final analysis cut-off date) | 0 | 0
Not Completed | 52 | 51
Not completed — Not treated | 2 | 0
Not completed — Covid-19 related | 1 | 1
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Adverse Event | 4 | 6
Not completed — Progressive disease | 37 | 31
Not completed — Study closure | 2 | 2
Not completed — Sponsor decision/recommendation | 3 | 2
Not completed — Switched to other drug/therapy | 2 | 2
Not completed — Lack of clinical benefit | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS): The randomised set included all randomised patients, regardless of whether they received treatment or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane | Placebo + 10 mg Everolimus + 25 mg Exemestane | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (11.3) | 60.3 (9.6) | 60.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 51 | 103
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 43 | 41 | 84
  Unknown or Not Reported | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 44 | 41 | 85
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) defined as the time from randomisation until progressive disease (PD) according to Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) in combination with modified MD Anderson Criteria (for bone lesion assessment), based on blinded independent assessment or death from any cause, whichever occurred earlier. As per RECIST, PD is defined as at least a 20% increase in the sum of diameters of target lesions, unequivocal progression of non-target lesions or the appearance of new lesions.
Time Frame: From randomisation until the earliest of disease progression, death or the time point of primary PFS analysis, up to 892 days.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane | Placebo + 10 mg Everolimus + 25 mg Exemestane
Number analyzed (Participants) | 52 | 51
Months | 12.7 [6.8 to 29.3] | 11.0 [7.7 to 19.5]
Statistical Analysis 1: Comparison: 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane vs Placebo + 10 mg Everolimus + 25 mg Exemestane; Cox proportional hazards model stratified for presence of baseline bone-only metastases, prior cyclin-dependent kinase (CDK) 4/6 inhibitor treatment and menopause status; Test type: Other; p = 0.6534, Log-rank test; Two-sided log-rank test stratified for presence of baseline bone-only metastases, prior (CDK) 4/6 inhibitor treatment and menopause status; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.55 to 2.59] — Comparison vs. Placebo+Everolimus+Exemestane

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) defined as the time from randomisation until death from any cause. For patients with 'event' as an outcome for OS:
  OS[days] = date of outcome - date of randomisation + 1.
  For patients with 'censored' as an outcome for OS:
  OS (censored)[days] = date of outcome - date of randomisation + 1.
Time Frame: From randomisation until death from any cause, up to 995 days.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane | Placebo + 10 mg Everolimus + 25 mg Exemestane
Number analyzed (Participants) | 52 | 51
Months | NA [22.3 to NA] — Median and upper bound of 95% CI could not be estimated due to insufficient events and data immaturity. | NA [22.3 to NA] — Median and upper bound of 95% CI could not be estimated due to insufficient events and data immaturity.
Statistical Analysis 1: Comparison: 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane vs Placebo + 10 mg Everolimus + 25 mg Exemestane; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.1797, Log rank test; Two-sided log-rank test stratified for presence of baseline bone-only metastases, prior CDK 4/6 inhibitor treatment and menopause status; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.18 to 1.40] — Comparison vs. Placebo+Everolimus+Exemestane

3. Secondary Outcome: Number of Patients With Disease Control (DC)
Description: Disease control (DC) was defined as a best overall response (BOR) of either complete response (CR), partial response (PR), stable disease (SD) or Non-CR/No-PD. SD and Non-CR/Non-PR must have been observed up until at least week 24 tumor assessment. BOR was defined according to RECIST v1.1 in combination with modified MD Anderson Criteria (for bone lesion assessment) based on all evaluable tumor assessments from randomisation until the earliest of PD, start of subsequent anti-cancer therapy, loss to follow-up, withdrawal of consent or death. To be aligned with the primary endpoint derivation, tumor assessments after two or more consecutively misses assessments were not considered. DC was assessed by independent reviewers.
Time Frame: From randomisation until the earliest of progressive disease or death from any cause, up to 892 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane | Placebo + 10 mg Everolimus + 25 mg Exemestane
Number analyzed (Participants) | 52 | 51
Participants | 29 | 25
Statistical Analysis 1: Comparison: 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane vs Placebo + 10 mg Everolimus + 25 mg Exemestane; Test type: Other; p = 0.4932, Regression, Logistic; Logistic regression model adjusted for presence of baseline bone-only metastases, prior CDK 4/6 inhibitor treatment and menopause status; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.60 to 2.86] — Comparison vs. Placebo+everolimus+exemestane. An odds ratio >1 indicates a benefit to the xentuzumab arm

4. Secondary Outcome: Duration of Disease Control (DC)
Description: Duration of disease control (DC), defined as the time from randomisation until the earliest of disease progression (according to Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) in combination with modified MD Anderson Criteria (for bone lesion assessment) or death from any cause, among patients with DC. Duration of DC was assessed by independent reviewers.
  The duration of DC was calculated as followed:
  For patients with disease progression or death:
  Duration of DC [days] = date of outcome - date of randomisation + 1
  For patients without disease progression or death:
  Duration of DC (censored) [days] = date of outcome - date of randomisation + 1
Time Frame: From randomisation until the earliest of progressive disease or death from any cause, up to 892 days.
Population: Randomised Set (RS): The randomised set included all randomised patients, regardless of whether they received treatment or not. Only participants with disease control are reported.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane | Placebo + 10 mg Everolimus + 25 mg Exemestane
Number analyzed (Participants) | 29 | 25
Months | 14.6 [9.2 to 29.3] | 18.4 [9.2 to NA] — Insufficient events to estimate upper bound of 95% CI for median.

5. Secondary Outcome: Number of Participants With Objective Response (OR)
Description: Number of participants with objective response (OR) by independent assessment. OR is defined as a best overall response of complete response (CR) or partial response (PR). Best overall response is defined according to RECIST v1.1 in combination with modified MD Anderson Criteria (for bone lesion assessment) and will consider all tumor assessments from randomisation until the earliest of PD, start of subsequent anti-cancer therapy, loss to follow-up, withdrawal of consent or death. To be aligned with the primary endpoint derivation, tumor assessments after two or more consecutively misses assessments were not considered.
Time Frame: From randomisation until end of treatment, up to 892 days.
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane | Placebo + 10 mg Everolimus + 25 mg Exemestane
Number analyzed (Participants) | 52 | 51
Participants | 6 | 5
Statistical Analysis 1: Comparison: 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane vs Placebo + 10 mg Everolimus + 25 mg Exemestane; Test type: Other; p = 0.7759, Regression, Logistic; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.20, 95% CI 2-sided [0.34 to 4.43] — Comparison vs. Placebo+everolimus+exemestane. An odds ratio >1 indicates a benefit to the xentuzumab arm

6. Secondary Outcome: Time to Pain Progression or Intensification of Pain Palliation
Description: Time to pain progression or intensification of pain palliation was defined as the time from randomisation until the earliest of:
  * 2 point increase from baseline in the Brief Pain Inventory - Short Form (BPI-SF), Item 3 (worst pain), without a decrease (of ≥1 point) from baseline analgesics use (via the 8-point Analgesic Quantification Algorithm [AQA]), or
  * 2 point increase from baseline in the AQA, or Death.
Time Frame: From randomisation until the earliest of pain progression, intensification of pain palliation, death or the time point of progression free survival analysis, up to 843 days.
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane | Placebo + 10 mg Everolimus + 25 mg Exemestane
Number analyzed (Participants) | 52 | 51
Months | 5.6 [3.2 to 9.3] | 3.0 [1.9 to NA] — Insufficient events to estimate upper bound of 95% CI for median.
Statistical Analysis 1: Comparison: 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane vs Placebo + 10 mg Everolimus + 25 mg Exemestane; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.9279, Log Rank; Two-sided log-rank test stratified for presence of baseline bone-only metastases, prior CDK4/6 inhibitor treatment and menopause status; Cox Proportional Hazard = 0.97, 95% CI 2-sided [0.54 to 1.76] — Comparison versus Placebo+everolimus+exemestane

ADVERSE EVENTS:
Time Frame: [All-cause mortality]: From signing informed consent until end of study, up to 1106 days. [Serious and other adverse events]: From first drug administration until end of treatment + 42 days of residual effect period, up to 939 days.
Description: [All-cause mortality]: Randomised Set (RS) including all randomised patients, regardless of whether they received treatment or not.
  [Serious and other adverse events]: Treated Set (TS) including all patients who are documented to have received and taken at least one dose of any study medication.
Arm/Group | 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane | Placebo + 10 mg Everolimus + 25 mg Exemestane
All-Cause Mortality (participants affected / at risk) | 6/52 | 10/51
Serious Adverse Events (participants affected / at risk) | 13/50 | 18/51
Other Adverse Events (participants affected / at risk) | 48/50 | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane (N=50) | Placebo + 10 mg Everolimus + 25 mg Exemestane (N=51)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Tongue abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 3 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Oophorectomy bilateral (Surgical and medical procedures) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1000 mg Xentuzumab + 10 mg Everolimus + 25 mg Exemestane (N=50) | Placebo + 10 mg Everolimus + 25 mg Exemestane (N=51)
Anaemia (Blood and lymphatic system disorders) | 10 | 13
Neutropenia (Blood and lymphatic system disorders) | 9 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 1
Ear pain (Ear and labyrinth disorders) | 3 | 0
Vertigo (Ear and labyrinth disorders) | 5 | 2
Dry eye (Eye disorders) | 5 | 3
Lacrimation increased (Eye disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Abdominal pain upper (Gastrointestinal disorders) | 7 | 4
Constipation (Gastrointestinal disorders) | 5 | 9
Diarrhoea (Gastrointestinal disorders) | 28 | 17
Dry mouth (Gastrointestinal disorders) | 5 | 8
Dyspepsia (Gastrointestinal disorders) | 4 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 18 | 14
Oral pain (Gastrointestinal disorders) | 3 | 1
Stomatitis (Gastrointestinal disorders) | 14 | 15
Toothache (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 9 | 8
Asthenia (General disorders) | 10 | 13
Chest pain (General disorders) | 3 | 4
Fatigue (General disorders) | 22 | 17
Influenza like illness (General disorders) | 5 | 3
Mucosal inflammation (General disorders) | 15 | 17
Oedema peripheral (General disorders) | 4 | 9
Pain (General disorders) | 3 | 5
Pyrexia (General disorders) | 7 | 9
COVID-19 (Infections and infestations) | 0 | 5
Cellulitis (Infections and infestations) | 1 | 4
Gingivitis (Infections and infestations) | 0 | 3
Oral candidiasis (Infections and infestations) | 0 | 3
Tooth abscess (Infections and infestations) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Urinary tract infection (Infections and infestations) | 9 | 9
Contusion (Injury, poisoning and procedural complications) | 7 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 2
Alanine aminotransferase increased (Investigations) | 8 | 7
Aspartate aminotransferase increased (Investigations) | 5 | 8
Blood albumin decreased (Investigations) | 3 | 0
Blood calcium decreased (Investigations) | 4 | 0
Blood cholesterol increased (Investigations) | 4 | 3
Blood creatine phosphokinase increased (Investigations) | 7 | 4
Blood creatinine increased (Investigations) | 5 | 3
Blood glucose increased (Investigations) | 4 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 7
Blood triglycerides increased (Investigations) | 4 | 0
Gamma-glutamyltransferase increased (Investigations) | 6 | 4
Glycosylated haemoglobin increased (Investigations) | 5 | 3
Lymphocyte count decreased (Investigations) | 3 | 2
Neutrophil count decreased (Investigations) | 4 | 6
Platelet count decreased (Investigations) | 9 | 5
Weight decreased (Investigations) | 7 | 5
White blood cell count decreased (Investigations) | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 18 | 18
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 13
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 5 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 8
Pain in jaw (Musculoskeletal and connective tissue disorders) | 3 | 1
Dizziness (Nervous system disorders) | 9 | 4
Dysgeusia (Nervous system disorders) | 10 | 6
Headache (Nervous system disorders) | 20 | 12
Paraesthesia (Nervous system disorders) | 6 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 2 | 5
Depression (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 7 | 5
Dysuria (Renal and urinary disorders) | 4 | 3
Pollakiuria (Renal and urinary disorders) | 4 | 2
Proteinuria (Renal and urinary disorders) | 1 | 3
Pelvic pain (Reproductive system and breast disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 8
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 6 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 9
Rash (Skin and subcutaneous tissue disorders) | 13 | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 3
Hypertension (Vascular disorders) | 6 | 8
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 4
Sciatica (Nervous system disorders) | 0 | 3
Glycosuria (Renal and urinary disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT03659136/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT03659136/SAP_001.pdf